CLINICAL TRIAL: NCT01733992
Title: A Phase 1, Single Center, Randomized, Double-Blind, Placebo-Controlled, Ascending Dose, Pharmacokinetics, Tolerability and Safety Study of R932348 Ophthalmic Solution in Patients With Mild to Moderate Keratoconjunctivitis Sicca
Brief Title: A Safety, Tolerability and Pharmacokinetics Study of R932348 Eye Drops in Patients With Dry Eye Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-932348-002
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Keratoconjunctivitis Sicca
MeSH Terms: conditions — Keratoconjunctivitis Sicca

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- R348 Ophthalmic Solution, 0.2% (Active Comparator): R348 Ophthalmic Solution, 0.2%, single (1 day) and multiple ascending dose (13 days) followed by a single dose on the fourteenth day.
  Interventions: Drug: R348 Ophthalmic Solution, 0.2%; Drug: Placebo
- R348 Ophthalmic Solution, 0.5% (Active Comparator): R348 Ophthalmic Solution, 0.5%, single (1 day) and multiple ascending dose (13 days) followed by a single dose on the fourteenth day.
  Interventions: Drug: R348 Ophthalmic Solution, 0.5%; Drug: Placebo
- R348 Ophthalmic Solution, 1.0% (Active Comparator): R348 Ophthalmic Solution, 1.0%, single (1 day) and multiple ascending dose (13 days) followed by a single dose on the fourteenth day.
  Interventions: Drug: R348 Ophthalmic Solution, 1.0%; Drug: Placebo
- Placebo (Placebo Comparator): Placebo, single (1 day) or multiple ascending dose (13 days) followed by a single dose on the fourteenth day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: R348 Ophthalmic Solution, 0.2% — R348 Ophthalmic Solution, 0.2% single and multiple ascending dose
  Other Names: R932348
  Arms: R348 Ophthalmic Solution, 0.2%
Drug: R348 Ophthalmic Solution, 0.5% — R348 Ophthalmic Solution, 0.5%, single and multiple ascending dose
  Other Names: R932348
  Arms: R348 Ophthalmic Solution, 0.5%
Drug: R348 Ophthalmic Solution, 1.0% — R348 Ophthalmic Solution, 1.0%, single and multiple ascending dose
  Other Names: R932348
  Arms: R348 Ophthalmic Solution, 1.0%
Drug: Placebo — Placebo, single and multiple ascending dose

SUMMARY:
The purpose of this study is to determine the safety, tolerability and pharmacokinetics of R348 eye drops in patients with dry eye disease.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled single and multiple ascending dose study to evaluate the ocular tolerability, safety, and pharmacokinetics of R348 administered in patients with mild to moderate keratoconjunctivitis sicca (KCS).

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate Keratoconjunctivitis Sicca.
* A corrected visual acuity in both eyes of 20/40 or better.
* An intraocular pressure of < 21 mm Hg with a difference between eyes of < 6 mm Hg.

Exclusion Criteria:

* History or evidence of ocular infection, inflammation, or conjunctivitis within 2 months prior to the first dosing day.
* History or evidence of blepharitis requiring the use of antibiotics or eye scrubs within 2 months prior to the first dosing day.
* History of herpes simplex keratitis at any time.
* Current ocular allergy symptoms.
* Recent use of eye medications such as steroids or cyclosporine
* Refractive eye surgery within 12 months of the first dosing day.
* Other eye surgeries within 4 months of the first dosing day.
* Current use of contact lenses or discontinuation of contact lens use within 2 weeks of the first dosing day.
* Receipt of any blood or blood products within 90 days prior to the first dosing day.
* Participation in any clinical study within 30 days prior to the first dosing day.
* History of disease, or currently have a significant illness or abnormal laboratory finding as determined by your study doctor.
* Positive for hepatitis B, hepatitis C or HIV.
* Smoked regularly within 12 months of first dosing day.
* History of substance abuse, drug addiction or alcoholism.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in corneal fluorescein staining | Baseline and Visits 4, 8 and 12

SECONDARY OUTCOMES:
Change in conjunctival lissamine green staining | Baseline and Visits 4, 8 and 12

OTHER OUTCOMES:
Change in Schirmer test | Baseline and Visits 4, 8 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Andover Eye Associates
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States